CLINICAL TRIAL: NCT05986617
Title: Wearable Bioimpedance Analyzer for Tracking Body Composition Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of feasibility due to study device issues.
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jacob M. Elkins, Assistant Professor of Orthopedics and Rehabilitation, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202207288
Record Dates: First submitted 2023-05-03; First posted 2023-08-14 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Knee Osteoarthritis
Keywords: total knee replacement; obesity; total joint replacement; bioimpedance; orthopedics; body composition; fitness tracker
MeSH Terms: conditions — Obesity; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Wearable Device Group (Experimental): Will be given InBody Band 2 to use while trying to achieve weight loss goal prior to total joint arthroplasty.
  Interventions: Device: InBody Band 2
- Control Group (No Intervention): Will not be given InBody Band 2 to use while trying to achieve weight loss goal prior to total joint arthroplasty.

INTERVENTIONS:
Device: InBody Band 2 — Wearable bioimpediance monitor similar to a fitness watch.
  Arms: Wearable Device Group

SUMMARY:
Obesity, namely at body mass index (BMI) levels exceeding 40kg/m2 (class III obesity), is a risk factor for many diseases including osteoarthritis (OA). In arthroplasty, patients in this population frequently present for and are turned away from surgical intervention. Subsequently, efforts are made to decrease BMI through simple weight loss, yet these have been suggested as ineffective and counterproductive. Furthermore, simple weight loss may include muscle mass loss, which is an additional risk factor for surgery. At the University of Iowa Hospitals and Clinics Orthopedics Department, efforts have been made to encourage muscle mass gain and body fat loss over simple weight loss where progress has been tracked through stationary, multi-frequency bioimpedance analysis (BIA). BIA is a readily available technology offered to industry and consumers, and BIA has recently been incorporated into wearable devices. In the UIHC Orthopedics department, a novel clinic aimed at holistically serving the osteoarthritic-class III obese population for controlled and monitored weight loss through BIA.

This study, a randomized controlled trial, aims to recruit adult patients with class III obesity presenting to the arthroplasty-obesity clinic. While all patients will receive individual body composition coaching to increase muscle mass and decrease body fat mass, they will be randomized to one of two cohorts: the study group will receive a wearable BIA wristband (InBody BAND 2) and instruction on its use in addition to the standard coaching, and the control group will only receive the standard coaching.

This study aims to identify if the use of a wearable BIA wristband aids in the desired body composition changes. In addition, this study aims to quantify the body composition changes exhibited by each cohort. Finally, this study aims to track surgical outcomes for those patients that are indicated for total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/= 18 years
* BMI > 40kg/m2
* Presenting to bariatric arthroplasty clinic with desire for total joint arthroplasty procedure
* Owns a smartphone capable of handling iOS or Google Play apps
* Has a wrist circumference less than or equal to 7.7"

Exclusion Criteria:

* Has a pacemaker or other electronic pacemaker placement
* Inability to complete study protocols
* Inability to stand unsupported for 60-90 seconds
* Does not own a smart phone capable of handling iOS or Google Play apps
* Has a wrist circumference greater than 7.7"

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Elkins, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Workgroup of the American Association of Hip and Knee Surgeons Evidence Based Committee. Obesity and total joint arthroplasty: a literature based review. J Arthroplasty. 2013 May;28(5):714-21. doi: 10.1016/j.arth.2013.02.011. Epub 2013 Mar 19. PMID 23518425
- [Background] Andrew JG, Palan J, Kurup HV, Gibson P, Murray DW, Beard DJ. Obesity in total hip replacement. J Bone Joint Surg Br. 2008 Apr;90(4):424-9. doi: 10.1302/0301-620X.90B4.20522. PMID 18378913
- [Background] DeMik DE, Bedard NA, Dowdle SB, Elkins JM, Brown TS, Gao Y, Callaghan JJ. Complications and Obesity in Arthroplasty-A Hip is Not a Knee. J Arthroplasty. 2018 Oct;33(10):3281-3287. doi: 10.1016/j.arth.2018.02.073. Epub 2018 Feb 26. PMID 29631859
- [Background] Foreman CW, Callaghan JJ, Brown TS, Elkins JM, Otero JE. Total Joint Arthroplasty in the Morbidly Obese: How Body Mass Index >/=40 Influences Patient Retention, Treatment Decisions, and Treatment Outcomes. J Arthroplasty. 2020 Jan;35(1):39-44. doi: 10.1016/j.arth.2019.08.019. Epub 2019 Aug 17. PMID 31530460
- [Background] Inacio MC, Kritz-Silverstein D, Raman R, Macera CA, Nichols JF, Shaffer RA, Fithian DC. The impact of pre-operative weight loss on incidence of surgical site infection and readmission rates after total joint arthroplasty. J Arthroplasty. 2014 Mar;29(3):458-64.e1. doi: 10.1016/j.arth.2013.07.030. Epub 2013 Sep 7. PMID 24018161
- [Background] Inacio MC, Kritz-Silverstein D, Raman R, Macera CA, Nichols JF, Shaffer RA, Fithian DC. The risk of surgical site infection and re-admission in obese patients undergoing total joint replacement who lose weight before surgery and keep it off post-operatively. Bone Joint J. 2014 May;96-B(5):629-35. doi: 10.1302/0301-620X.96B5.33136. PMID 24788497
- [Background] Friedman RJ, Hess S, Berkowitz SD, Homering M. Complication rates after hip or knee arthroplasty in morbidly obese patients. Clin Orthop Relat Res. 2013 Oct;471(10):3358-66. doi: 10.1007/s11999-013-3049-9. Epub 2013 May 14. PMID 23670675
- [Background] Ward LC, Dyer JM, Byrne NM, Sharpe KK, Hills AP. Validation of a three-frequency bioimpedance spectroscopic method for body composition analysis. Nutrition. 2007 Sep;23(9):657-64. doi: 10.1016/j.nut.2007.06.009. PMID 17679047
- [Background] Milone MT, Shenoy K, Pham H, Jazrawi LM, Strauss EJ. MRI analysis of peripheral soft tissue composition, not body mass index, correlates with outcomes following anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2018 Dec;26(12):3711-3716. doi: 10.1007/s00167-018-4966-7. Epub 2018 May 3. PMID 29725746
- [Background] Muller M, Tohtz S, Winkler T, Dewey M, Springer I, Perka C. MRI findings of gluteus minimus muscle damage in primary total hip arthroplasty and the influence on clinical outcome. Arch Orthop Trauma Surg. 2010 Jul;130(7):927-35. doi: 10.1007/s00402-010-1085-4. Epub 2010 Mar 11. PMID 20221834
- [Background] Pichonnaz C, Bassin JP, Currat D, Martin E, Jolles BM. Bioimpedance for oedema evaluation after total knee arthroplasty. Physiother Res Int. 2013 Sep;18(3):140-7. doi: 10.1002/pri.1540. Epub 2012 Nov 27. PMID 23188719
- [Background] Qin ES, Bowen MJ, James SL, Chen WF. Multi-segment bioimpedance can assess patients with bilateral lymphedema. J Plast Reconstr Aesthet Surg. 2020 Feb;73(2):328-336. doi: 10.1016/j.bjps.2019.06.041. Epub 2019 Aug 7. PMID 31515193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period dates: 07/14/2023 - 05/31/2024 Types of location: medical clinic
Period: Overall Study
Arm/Group | Wearable Device Group | Control Group
Started | 30 | 30
Completed | 1 | 5
Not Completed | 29 | 25

BASELINE CHARACTERISTICS:
Population: Not different from assignment in participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wearable Device Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 15 | 45
  >=65 years | 0 | 15 | 15
Age, Continuous [Mean (Full Range); unit: years] | 57.6 [35 to 77] | 58.1 [43 to 81] | 57.9 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Body mass index (BMI) [Mean (Full Range); unit: units on a scale (kg/m^2)] | 49.8 [42.7 to 59.0] | 50.9 [41.8 to 65.9] | 50.3 [41.8 to 65.9]

OUTCOME MEASURES:

1. Primary Outcome: Device Impact on Length of Time Until Surgical Indication
Description: In this RCT, we analyzed the impact of the wearable device (band) on length of time until surgical indication
Time Frame: Maximum 12 months prior to TJA
Population: 6 total subjects were indicated for surgery. 3 per group.
Measure: Mean (Full Range); unit: months
Arm/Group | Wearable Device Group | Control Group
Number analyzed (Participants) | 3 | 3
months | 3.7 [3 to 7] | 8.7 [7 to 10]
Statistical Analysis 1: Comparison: Wearable Device Group vs Control Group; Power calculation: 2 factor (group, time) ANOVA design with a group*time interaction term to estimate the proposed sample size. Using a Cohen's effect size estimate for 2 groups with 5 time-points, a sample size of 40 per group will provide >90% to detect a moderate effect size (0.25) for group, for time and for the group*time interaction; Test type: Superiority; p = .06429, t-test, 2 sided — 2-tail t-test with non-equivalent variances

2. Secondary Outcome: Surgical Outcomes
Description: Incidence of complications in surgical outcomes for patients across both groups that achieve obtaining surgical indication.
Time Frame: 24 months postoperatively
Reporting Status: Not Posted

3. Secondary Outcome: Body Composition Changes Quantified
Description: Body mass change, fat mass change, skeletal muscle mass change
Time Frame: Maximum 12 months prior to TJA
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Wearable Device Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wearable Device Group (N=30) | Control Group (N=30)
Band Tightness Resulting in Wrist Pain and Ball on Wrist (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT05986617/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05986617/ICF_001.pdf